CLINICAL TRIAL: NCT03788057
Title: Evaluation of the Usefulness of Induced Sputum Eosinophilia, eNO and Bronchial Hyperresponsiveness in Predicting the Failure of Inhaled Corticosteroids Dose Reduction in Children and Adolescents With Stable Asthma
Brief Title: Inflammatory Indices in Predicting the Failure of Inhaled Corticosteroids Reduction in Young Participants With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute for Tuberculosis and Lung Diseases, Poland (Other)
Collaborators: University of Rzeszow (Other); The Regional Public Hospital in Lesko, Poland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NITLD
Record Dates: First submitted 2018-12-12; First posted 2018-12-27 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2018-12

CONDITIONS: Asthma Chronic

STUDY DESIGN:
Intervention Model Description: A prospective, observational, interventional, single blind study. Clinician takes decision about possible reduction of ICS dose basing on clinical data only - is not aware of the results of the inflammatory parameters measurement.
Masking Description: Clinician takes decision about possible change in treatment basing on clinical data only - is not aware of the results of the inflammatory parameters measurements
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- stable asthma (Other): In patients with previously stable course of the asthma, every 3 months the symptoms are evaluated and the dose of ICS is customized - in accordance with the GINA guidelines. This decision is based solely on clinical data (control of symptoms) and is the same as in patients not participating in the study.
  In patients participating in the study, inflammatory parameters are also measured (sputum eosinophilia, eNO, EBT, bronchial reactivity), but results are not known to clinician taking decision about possible ICS dose reduction.
  Interventions: Other: ICS dose reduction

INTERVENTIONS:
Other: ICS dose reduction — If control of symptoms is maintained (evaluation based on clinical symptoms solely), every 3 months the dose of ICS is halved according to GINA guidelines, until the control is lost or the lowest daily dose is reached (200 mcg, calculated as budesonide equivalent).
  In the case of loss of asthma control, beta-mimetic will be administered (temporarily) and return to the chronic administration of the previous, twice higher dose of ICS is restored (or further increase of treatment). In severe exacerbations, inclusion of oral steroids will be considered.

SUMMARY:
A prospective, observational, interventional, single-blind study (blinded for a clinician in the field of inflammatory parameters).

The aim of the study is evaluation of the usefulness of induced sputum eosinophilia and other inflammatory indices [exhaled nitric oxide (NO), exhaled breath temperature, bronchial hyperresponsiveness] in predicting the failure of treatment reduction with inhaled corticosteroids (ICS) in stable asthma in children and adolescents.

In participants with a stable course of the asthma (confirmed in the run -in period), every 3 months the dose of ICS is halved (according to GINA guidelines) until the control is lost or the lowest daily ICS dose is reached (200 mcg, calculated as budesonide equivalent). Throughout the treatment reduction period, the participants run an observation card (clinical symptoms) and peak expiratory flow rate (PEFR) measurements. Clinical evaluation is performed every month, with spirometry, exhaled NO and exhaled breath temperature measurements. Before the reduction and then one month after the change of treatment, the hyperresponsiveness measurement is carried out with the sputum induction (combined method using hypertonic saline), and 2 months after the change of treatment with the exercise challenge test.

In the case of loss of asthma control, beta-mimetic will be administered (temporarily) and return to dose of ICS before reduction or further increase of treatment is planned. In severe asthma exacerbations, oral steroids will be considered.

The study is observational: treatment is modified according to GINA guidelines based on clinical data as part of routine medical care. Only difference compared do standard care is supplementary inflammation evaluation (exhaled NO, sputum eosinophilia, bronchial hyperreactivity).

DETAILED DESCRIPTION:
Introduction Guidelines for the treatment of asthma recommend the use of the smallest dose of inhaled steroid (ICS), which allows to maintain control of the symptoms of the disease. The GINA 2006 guidelines proposed (and later editions it upheld) that in the case of symptom control by monotherapy with ICS, to reduce their dose every 3 months, up to the lowest dose administered once a day, which should be used for one year before taking possible decision to stop it.

There are no clear of simple and sensitive indicators that would allow detection of a threatening loss of control before the clinical symptoms worsen.

Aim of the study Evaluation of the usefulness of induced sputum eosinophilia and other inflammatory indices [exhaled nitric oxide (NO), exhaled breath temperature (EBT), bronchial hyperresponsiveness] in predicting the failure of treatment reduction with inhaled corticosteroids in stable asthma in children and adolescents.

Subjects Participants aged 12-18 years with stable asthma (mild or moderate), treated in the Allergy Clinic of the Hospital in Lesko with medium doses in ICS. The severity of asthma was initially determined in accordance with the GINA criteria and verified during several years of observation by the assessment of clinical symptoms, functional examinations and the dose of inhaled steroids controlling the disease.

Project description A prospective, observational, single-blind study (blinded for a clinician in the field of inflammatory parameters). Clinician takes decision about possible reduction of ICS dose basing on clinical data only - is not aware of the results of the inflammatory parameters measurement.

The study is consisting of two periods:

First period (run - in):

A four-week run - in period in which clinical symptoms and the use of short acting beta2 agonists (SABA) and PEFR are monitored. At the end of this period, in participants with stable disease the following parameters are measured: eNO, EBT, spirometry, and sputum induction with hyperosmolar saline in combination with the hyperresponsiveness. Before the reduction of treatment on another day, an exercise challenge test is also performed.

The criteria for the stability of asthma in the run - in period are:

* symptoms no more than 3 times a week
* SABA use less than 3 times a week
* without night wake up
* PEFR variability below 20%
* FEV1 above 80% of predicted

Second period of the study - reduction of anti-inflammatory therapy. In participants with previously stable course of the asthma (confirmed in the run -in period), the control of asthma is monitored regularly throughout the observation period. All participants run an observation card (clinical symptoms) and PEFR measurements. Monthly spirometry, exhaled NO and exhaled breath temperature measurements are performed. Every 3 months and one month after the change of treatment (i.e in months 0, 1, 3, 4, 6 and 7), the hyperresponsiveness measurement is carried out with the sputum induction (combined method, [7]). Two months after the dose change (months 2, 5, 8) the exercise challenge test is carried out.

Every 3 months control of the asthma symptoms is evaluated taking account the clinical data, and possible change of ICS dose is considered. Results of bronchial reactivity measurements and sputum cytology are not known to clinician who decide on a possible ICS dose change - he is blinded to the results of tests and the therapeutic decision is based solely on clinical evaluation.

In participants with a stable course of the disease over past 3 months, the dose of ICS is halved, in accordance with GINA guidelines. In the case of loss of asthma control, appropriate treatment modifications are administered and the patient is withdrawn from the study.

Participation in the study is continued until asthma control is lost or the lowest daily dose is reached (200 mcg, calculated as budesonide equivalent) - without losing asthma control at next visit.

Measurements

1. Daily clinical evaluation by the patient:

   * symptoms score according to the Santanello questionnaire
   * PEFR measurement
2. Every month

   * Asthma Control Test
   * spirometry [forced expiratory flow in 1st second (FEV1), forced vital capacity (FVC), forced expiratory flow between 25% and 75% of FVC (FEF25-75)]
   * eNO measurement
   * exhaled breath temperature measurement (EBT)
3. every 3 months

   * quality of life test (QoL, Polish version of the questionnaire), i.e. months 3, 6, 9
   * cytological evaluation of induced sputum (i.e. months 0, 1, 3, 4, 6, 7)
   * assessment of bronchial hyperresponsiveness:

     * one month after the ICS dose reduction and then before each subsequent dose reduction in ICS ((i.e. months 0, 1, 3, 4, 6, 7) - during the sputum induction with hyperosmolar salt (combined method)
     * 2 months after each treatment reduction (i.e. months 2, 5, 8): exercise challenge test (6-minute free-running test monitored by pulse)

Criteria for loss of control [1, 6] - any of the following:

* use of bronchodilators> 5 times a week
* the need for treatment with oral corticosteroids
* PEFR decrease above 20% for 2 consecutive days, compared to the average run-in period In the case of loss of asthma control, beta-mimetic will be administered (temporarily) and return to the chronic administration of the previous, twice higher dose of ICS is restored (or further increase of treatment). In severe exacerbations, inclusion of oral steroids will be considered.

Criteria for discontinuation of participation in the study

1. Loss of asthma control (treatment strategy: beta-mimetic temporarily, return to dose of ICS before reduction or further increase of treatment; in severe exacerbations, inclusion of oral steroids).
2. Lack of adherence to the recommendations or failure to report.

The staff of the center has experience in the production of sputum induction in participants with asthma [Ciółkowski J, Mazurek H, Stasiowska B. Evaluation of step - down therapy from an inhaled steroid to montelukast in childhood asthma. Allergologia et immunopathologia (Madr.), 2014: Jul - Aug; 42 (4): 282 - 288].

The test will be performed in conditions ensuring patient safety, with the availability of an anaesthesiologist and anti-shock kit.

ELIGIBILITY:
Inclusion Criteria:

* mild or moderate asthma with a stable course of at least 3 months:

  * symptoms less than 4x per week,
  * use of SABA below 3x a week,
  * night awakening below 1x per week,
  * FEV1> 80% of predicted
  * no dose change in ICS or use of systemic steroids from 3 months
* good adherence to treatment

Exclusion Criteria:

* infection or exacerbation of asthma requiring the use of systemic steroids (or changes in the dose of inhaled steroids) in the last 3 months before the study
* other chronic lung diseases or general diseases affecting the respiratory system
* tobacco smoking
* FEV1 below 80% of the predicted value

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Regional Public Hospital in Lesko, Poland, Lesko, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] www.ginasthma.org
- [Result] Zacharasiewicz A, Wilson N, Lex C, Erin EM, Li AM, Hansel T, Khan M, Bush A. Clinical use of noninvasive measurements of airway inflammation in steroid reduction in children. Am J Respir Crit Care Med. 2005 May 15;171(10):1077-82. doi: 10.1164/rccm.200409-1242OC. Epub 2005 Feb 11. PMID 15709050
- [Result] Green RH, Brightling CE, McKenna S, Hargadon B, Parker D, Bradding P, Wardlaw AJ, Pavord ID. Asthma exacerbations and sputum eosinophil counts: a randomised controlled trial. Lancet. 2002 Nov 30;360(9347):1715-21. doi: 10.1016/S0140-6736(02)11679-5. PMID 12480423
- [Result] Fleming L, Wilson N, Regamey N, Bush A. Use of sputum eosinophil counts to guide management in children with severe asthma. Thorax. 2012 Mar;67(3):193-8. doi: 10.1136/thx.2010.156836. Epub 2011 Aug 8. PMID 21825081
- [Result] Jayaram L, Pizzichini MM, Cook RJ, Boulet LP, Lemiere C, Pizzichini E, Cartier A, Hussack P, Goldsmith CH, Laviolette M, Parameswaran K, Hargreave FE. Determining asthma treatment by monitoring sputum cell counts: effect on exacerbations. Eur Respir J. 2006 Mar;27(3):483-94. doi: 10.1183/09031936.06.00137704. PMID 16507847
- [Result] Li AM, Tsang TW, Lam HS, Sung RY, Chang AB. Predictors for failed dose reduction of inhaled corticosteroids in childhood asthma. Respirology. 2008 May;13(3):400-7. doi: 10.1111/j.1440-1843.2007.01222.x. PMID 18399863
- [Result] Prieto L, Bruno L, Gutierrez V, Uixera S, Perez-Frances C, Lanuza A, Ferrer A. Airway responsiveness to adenosine 5'-monophosphate and exhaled nitric oxide measurements: predictive value as markers for reducing the dose of inhaled corticosteroids in asthmatic subjects. Chest. 2003 Oct;124(4):1325-33. doi: 10.1378/chest.124.4.1325. PMID 14555562
- [Result] Deykin A, Lazarus SC, Fahy JV, Wechsler ME, Boushey HA, Chinchilli VM, Craig TJ, Dimango E, Kraft M, Leone F, Lemanske RF, Martin RJ, Pesola GR, Peters SP, Sorkness CA, Szefler SJ, Israel E; Asthma Clinical Research Network, National Heart, Lung, and Blood Institute/NIH. Sputum eosinophil counts predict asthma control after discontinuation of inhaled corticosteroids. J Allergy Clin Immunol. 2005 Apr;115(4):720-7. doi: 10.1016/j.jaci.2004.12.1129. PMID 15805990
- [Result] Belda J, Parameswaran K, Lemiere C, Kamada D, O'Byrne PM, Hargreave FE. Predictors of loss of asthma control induced by corticosteroid withdrawal. Can Respir J. 2006 Apr;13(3):129-33. doi: 10.1155/2006/189127. PMID 16642226
- [Result] Jatakanon A, Lim S, Barnes PJ. Changes in sputum eosinophils predict loss of asthma control. Am J Respir Crit Care Med. 2000 Jan;161(1):64-72. doi: 10.1164/ajrccm.161.1.9809100. PMID 10619799
- [Result] Leuppi JD, Salome CM, Jenkins CR, Anderson SD, Xuan W, Marks GB, Koskela H, Brannan JD, Freed R, Andersson M, Chan HK, Woolcock AJ. Predictive markers of asthma exacerbation during stepwise dose reduction of inhaled corticosteroids. Am J Respir Crit Care Med. 2001 Feb;163(2):406-12. doi: 10.1164/ajrccm.163.2.9912091. PMID 11179114
- [Result] Cabral AL, Vollmer WM, Barbirotto RM, Martins MA. Exhaled nitric oxide as a predictor of exacerbation in children with moderate-to-severe asthma: a prospective, 5-month study. Ann Allergy Asthma Immunol. 2009 Sep;103(3):206-11. doi: 10.1016/S1081-1206(10)60183-4. PMID 19788017

RESULTS

PARTICIPANT FLOW:
Groups:
- Stable Asthma: In patients with previously stable course of the asthma, every 3 months the symptoms are evaluated and the dose of ICS is customized - in accordance with the GINA guidelines. This decision is based solely on clinical data (control of symptoms) and is the same as in patients not participating in the study.
  In patients participating in the study, inflammatory parameters are also measured (sputum eosinophilia, eNO, EBT, bronchial reactivity), but results are not known to clinician taking decision about possible ICS dose reduction.
  ICS dose reduction: If control of symptoms is maintained (evaluation based on clinical symptoms solely), every 3 months the dose of ICS is halved according to GINA guidelines, until the control is lost or the lowest daily dose is reached (200 mcg, calculated as budesonide equivalent).
  In the case of loss of asthma control, beta-mimetic will be administered (temporarily) and return to the chronic administration of the previous, twice higher dose of ICS is restored (or further increase of treatment). In severe exacerbations, inclusion of oral steroids will be considered.
Period: Overall Study
Arm/Group | Stable Asthma
Started | 58
Completed | 52
Not Completed | 6

BASELINE CHARACTERISTICS:
Groups:
- Stable Asthma: In patients with a previously stable course of asthma, every 3 months the symptoms are evaluated and the dose of ICS is customized - in accordance with the GINA guidelines. This decision is based solely on clinical data (control of symptoms) and is the same as in patients not participating in the study.
  In patients participating in the study, inflammatory parameters are also measured (sputum eosinophilia, eNO, EBT, bronchial reactivity), but results are not known to clinician taking decisions about possible ICS dose reduction.
  If control of symptoms is maintained (evaluation based on clinical symptoms solely), every 3 months the dose of ICS is halved according to GINA guidelines, until the control is lost or the lowest daily dose is reached (200 mcg, calculated as budesonide equivalent).
  Case of loss of asthma control: beta-mimetic will be administered (temporarily) and return to the chronic administration of the previous, twice higher dose of ICS is restored (or further increase of
Arm/Group | Stable Asthma
Number analyzed (Participants) | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 52
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 52
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients With Loss of Asthma Control
Description: Criteria for loss of control (any of the following):
  * use of bronchodilators > 5 times a week
  * the need for treatment with oral corticosteroids
  * PEFR decrease >20% for 2 consecutive days, compared to the average run-in period
Time Frame: at 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Stable Asthma
Number analyzed (Participants) | 52
Participants | 17

2. Secondary Outcome: Change in Sputum Eosinophilia
Description: eosinophil percentage in induced sputum compared to baseline
Time Frame: at 1, 3, 4, 6 and 7 month
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Change in Airway Hyperresponsiveness to Hypertonic Saline
Description: Airway hyperresponsiveness to hypertonic saline measured using combined method (together with sputum induction) and compared to baseline
Time Frame: at 1, 3, 4, 6 and 7 month
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Change in Airway Hyperresponsiveness (Exercise)
Description: Airway hyperresponsiveness measured using an exercise challenge test and compared to baseline
Time Frame: at 2, 5 and 8 month
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Change in Exhaled NO
Description: Measured every month and compared to baseline
Time Frame: months 1 - 8
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Change in Exhaled Breath Temperature (EBT)
Description: Measured every month and compared to baseline
Time Frame: months 1 - 8
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in FEV1
Description: Measured every month and compared to baseline
Time Frame: months 1 - 8
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in FVC
Description: Measured every month and compared to baseline
Time Frame: months 1 - 8
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in FEF25-75
Description: Measured every month and compared to baseline
Time Frame: months 1 - 8
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: During all the study period (1,5 year)
Arm/Group | Stable Asthma
All-Cause Mortality (participants affected / at risk) | 0/58
Serious Adverse Events (participants affected / at risk) | 0/58
Other Adverse Events (participants affected / at risk) | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-12-25): https://cdn.clinicaltrials.gov/large-docs/57/NCT03788057/Prot_000.pdf